CLINICAL TRIAL: NCT07354048
Title: Impact Of Thyroid Dysfunction on Liver Function Tests In Sohag University Hospital
Brief Title: Impact Of Thyroid Dysfunction on Liver Function Tests
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Omnia Ahmed Mohamed Aref, Resident, Internal Medicine Department, Faculty of Medicine, Sohag University, Sohag University
Other Study IDs: Soh-Med--25-7-9MS
Record Dates: First submitted 2025-09-30; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Disease
MeSH Terms: conditions — Thyroid Diseases | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group
  Interventions: Other: Control group
- Patients with hypothyroidism or hyperthyroidism that are controlled on treatment
  Interventions: Other: Patients with hypothyroidism or hyperthyroidism that are controlled on treatment
- Patients with hypothyroidism or hyperthyroidism that are not controlled on treatment
  Interventions: Other: Patients with hypothyroidism or hyperthyroidism that are not controlled on treatment
- Patients with hypothyroidism or hyperthyroidism that are firstly discovered
  Interventions: Other: Patients with hypothyroidism or hyperthyroidism that are firstly discovered

INTERVENTIONS:
Other: Control group — Healthy people
  Groups: Control group
Other: Patients with hypothyroidism or hyperthyroidism that are controlled on treatment — This group includes patients with hypothyroidism or hyperthyroidism that are controlled on treatment
  Groups: Patients with hypothyroidism or hyperthyroidism that are controlled on treatment
Other: Patients with hypothyroidism or hyperthyroidism that are not controlled on treatment — This group includes patients with hypothyroidism or hyperthyroidism that are not controlled on treatment
  Groups: Patients with hypothyroidism or hyperthyroidism that are not controlled on treatment
Other: Patients with hypothyroidism or hyperthyroidism that are firstly discovered — This group includes patients with hypothyroidism or hyperthyroidism that are firstly discovered
  Groups: Patients with hypothyroidism or hyperthyroidism that are firstly discovered

SUMMARY:
This study aims to evaluate the effect of thyroid dysfunction on liver function tests.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 20-60 years old either with Hypothyroidism or Hyperthyroidism (controlled on treatment or not) and firstly diagnosed Hypothyroidism or Hyperthyroidism.
* Euthyroid controls (clinically healthy control subjects were recruited from the general population with the same socio-economic status with the subjects.)

Exclusion Criteria:

* Patients aged < 20 years old.
* Patients With Liver Disease.
* Pregnant and lactating women.
* Patients with severe infections or sepsis.
* Patients with Heart Disease.
* Patients who on drugs that can affect liver function such as phenothiazine, phenylbutazone, methyldopa, among others.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients between the ages of 20-60 years old either with Hypothyroidism or Hyperthyroidism (controlled on treatment or not) and firstly diagnosed Hypothyroidism or Hyperthyroidism.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Measuring total bilirubin level in patients with thyroid dysfunction diseases | 1 months
  Collecting blood samples from the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Boelaert K, Franklyn JA. Thyroid hormone in health and disease. J Endocrinol. 2005 Oct;187(1):1-15. doi: 10.1677/joe.1.06131. PMID 16214936
- [Background] Malik R, Hodgson H. The relationship between the thyroid gland and the liver. QJM. 2002 Sep;95(9):559-69. doi: 10.1093/qjmed/95.9.559. PMID 12205333
- [Background] Bianco AC, Salvatore D, Gereben B, Berry MJ, Larsen PR. Biochemistry, cellular and molecular biology, and physiological roles of the iodothyronine selenodeiodinases. Endocr Rev. 2002 Feb;23(1):38-89. doi: 10.1210/edrv.23.1.0455. PMID 11844744